CLINICAL TRIAL: NCT02853955
Title: MitraClip® for the Treatment of Recurrent Severe Mitral Regurgitation After Surgical Mitral Valve Repair
Brief Title: MitraClip® After Surgical Mitral Valve Repair
Acronym: MVRepair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Daniel Braun, MD, MD, LMU Klinikum
Other Study IDs: GE IDE MucS001-16
Record Dates: First submitted 2016-03-31; First posted 2016-08-03 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Percutaneous edge-to-edge repair of the mitral valve — MitraClip in patients with recurrent MI after surgical mitral valve repair.

SUMMARY:
Percutaneous edge-to-edge repair of the mitral valve has been shown to be a safe and effective alternative treatment option for selected patients at high risk for cardiac surgery. Patients with recurrent mitral regurgitation after surgical mitral valve repair (sMVR) are per se at increased risk for another cardiac surgery. The purpose of this multicenter retrospective analysis of patients treated with a MitraClip® after sMVR, is to evaluate the effectiveness and durability of this minimally invasive treatment option in this subset of patients.

DETAILED DESCRIPTION:
In this multicenter retrospective analysis of MitraClip® cases after MVR the effectiveness and durability of this minimally invasive treatment option in this subset of patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients with recurrent mitral regurgitation treated with a MitraClip®.

Exclusion Criteria:

* Patient with endocarditis,
* Patients with torn mitral valve ring.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with a MitraClip® after sMVR
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
MR (mitral regurgitation) grade after clip treatment | 1 year
  Scale 0-4

SECONDARY OUTCOMES:
MR (mitral regurgitation) grade at latest follow up | 1 year
  Scale 0-4
NYHA status at latest follow up | 1 year
Distance in 6 minute walk test at latest follow up | 1 year
LVEF (left ventricular ejection fraction) at latest follow up | 1 year
LVEDV (left ventricular enddiastolic volume) at latest follow up | 1 year
LVEDD (lef ventricular enddiastolic diameter) at latest follow up | 1 year
Mean mitral valve gradient | 1 year
Procedural complications | index procedure
Death, recurrent mitral regurgitation grade > 2, repeat intervention/operation of mitral valve | 1 year
  combined endpoint defined as freedom from each Event (death, MR grade >2 or reintervention/Operation)
Clip success based on type of sMVR | index procedure
  success defined as reduction of 1 MR grade (scale 0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Hausleiter, MD, Study Chair — LMU Munich
Locations (1):
- Munich University Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No